CLINICAL TRIAL: NCT05022927
Title: A PHASE I STUDY OF ERY974 IN PATIENTS WITH LOCALLY ADVANCED OR METASTATIC HEPATOCELLULAR CARCINOMA
Brief Title: A Phase I Study of ERY974 in Patients With Hepatocellular Carcinoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERY103JG
Record Dates: First submitted 2021-06-28; First posted 2021-08-26 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — bispecific antibody ERY974; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose escalation part (Experimental): Patients will receive ERY974 in combination with atezolizumab and bevacizumab after administering ERY974 as a single agent and to determine the MTD by evaluating DLTs of in patients with locally advanced or metastatic HCC.
  Interventions: Drug: ERY974; Drug: Tocilicumab; Drug: Atezolizumab; Drug: Bevacizumab
- Expansion part (Experimental): Patients will receive ERY974 in combination with atezolizumab and bevacizumab after administering ERY974 as a single agent To evaluate the anti-tumor effect.
  Interventions: Drug: ERY974; Drug: Tocilicumab; Drug: Atezolizumab; Drug: Bevacizumab
- Concomitant use part (Experimental): Patients will receive ERY974 in combination with atezolizumab and bevacizumab and to determine the MTD.
  Interventions: Drug: ERY974; Drug: Tocilicumab; Drug: Atezolizumab; Drug: Bevacizumab
- Biomarker part (Experimental): Patients will receive ERY974 in combination with atezolizumab and bevacizumab after administering ERY974 as a single agent and to evaluate the biomarkers.
  Interventions: Drug: ERY974; Drug: Tocilicumab; Drug: Atezolizumab; Drug: Bevacizumab
- Mono dose escalation part (Experimental): Patients will receive ERY974 as a single agent and to determine the MTD by evaluating DLTs of in patients with locally advanced or metastatic HCC.
  Interventions: Drug: ERY974; Drug: Tocilicumab; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: ERY974 — ERY974 vial
Drug: Tocilicumab — Tocilizumab vial
Drug: Atezolizumab — Atezolizumab vial
Drug: Bevacizumab — Bevacizumab vial

SUMMARY:
This is a multicenter, open-label, dose-escalation study designed to determine the maximum tolerated dose (MTD) by evaluating dose-limiting toxicities (DLTs) and to evaluate the safety, tolerability, pharmacokinetics, anti-tumor effect, and biomarkers of ERY974 in combination with atezolizumab and bevacizumab following premedication with tocilizumab in patients with locally advanced or metastatic HCC.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years at time of informed consent
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) of 0 or 1
* HCC that has been histologically confirmed

Exclusion Criteria:

* Previous or concomitant autoimmune disease
* Uncontrolled diabetes mellitus and hypertension
* Concurrent New York Heart Association (NYHA) Class ≥II congestive heart failure, myocardial infarction, arrhythmia, or unstable angina, or a history thereof within 6 months before enrollment.
* Concurrent symptomatic cerebrovascular disorder (e.g., subarachnoid hemorrhage, cerebral infarction, or transient ischemic attack), or a history thereof within 6 months before enrollment.
* Symptomatic, untreated, or actively progressing CNS metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab (Dose limiting toxicities) [Dose escalation part] | At the end of Cycle 2 (Cycle 1 is 14day, Cycle 2 or later is 21days)
  Incidence and nature of DLTs
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab (Electrocardiograms in triplicate) [Dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab (Electrocardiograms in triplicate) [Dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Uncorrected QT interval, QTcF, PR duration, QRS interval and RR interval
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab (Electrocardiograms in triplicate) [Dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Heart Rate
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Maximum plasma concentration (Cmax) of ERY974 Maximum plasma concentration (Cmax) of ERY974 Maximum plasma concentration (Cmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Time to reach maximum plasma drug concentration (Tmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Area under the concentration versus time curve (AUC) of ERY974
Anti-tumor activity of ERY974 in combination with atezolizumab and bevacizumab [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Objective Response Rate (ORR) is defined as proportion of patients who had a confirmed complete response (CR) or partial response (PR), as determined by the investigator with use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab from initiation (Dose limiting toxicities) [Concomitant use part] | At the end of Cycle 1 (each Cycle is 21days)
  Incidence and nature of DLTs
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab (Adverse Events) [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab from initiation [Concomitant use part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Uncorrected QT interval, QTcF, PR duration, QRS interval and RR interval
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab from initiation [Concomitant use part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Heart Rate
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab from initiation [Concomitant use part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Maximum plasma concentration (Cmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab from initiation [Concomitant use part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Time to reach maximum plasma drug concentration (Tmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab from initiation [Concomitant use part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Area under the concentration versus time curve (AUC) of ERY974
Biomarkers of ERY974 in combination with atezolizumab and bevacizumab [Biomarker part] | From screening to 6weeks
  GPC3 and PD-L1 IHC staining
Biomarkers of ERY974 in combination with atezolizumab and bevacizumab [Biomarker part] | From screening to 6weeks
  Immune-related molecule IHC
Biomarkers of ERY974 in combination with atezolizumab and bevacizumab [Biomarker part] | From screening to 6weeks
  Gene expression
Anti-tumor activity of ERY974 [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Objective Response Rate (ORR) is defined as proportion of patients who had a confirmed complete response (CR) or partial response (PR), as determined by the investigator with use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Safety of ERY974 (Dose limiting toxicities) [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Incidence and nature of DLTs
Safety of ERY974 (Dose limiting toxicities) [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0
Safety of ERY974 (Dose limiting toxicities) [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Uncorrected QT interval, QTcF, PR duration, QRS interval and RR interval
Safety of ERY974 (Dose limiting toxicities) [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Heart Rate

SECONDARY OUTCOMES:
Anti-tumor activity of ERY974 in combination with atezolizumab and bevacizumab [Dose escalation part] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to about 52 weeks.
  Objective Response Rate (ORR) is defined as proportion of patients who had a confirmed complete response (CR) or partial response (PR), as determined by the investigator with use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Safety and tolerability of ERY974 in combination with atezolizumab and bevacizumab (Adverse Events) [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0
Safety, tolerability and pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab (Adverse Events) [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Uncorrected QT interval, QTcF, PR duration, QRS interval and RR interval
Safety, tolerability and pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab (Adverse Events) [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Heart Rate
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Maximum plasma concentration (Cmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Time to reach maximum plasma drug concentration (Tmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Area under the concentration versus time curve (AUC) of ERY974
Anti-tumor activity of ERY974 in combination with atezolizumab and bevacizumab from initiation [Concomitant use part] | From screening until disease progression, study discontinuation, withdrawal or death, whichever occurs first, assessed up to about 52 weeks.
  Objective Response Rate (ORR) is defined as proportion of patients who had a confirmed complete response (CR) or partial response (PR), as determined by the investigator with use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Safety of ERY974 in combination with atezolizumab and bevacizumab (Adverse Events) [Expansion part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Incidence, nature, and severity of adverse events (AEs) as assessed by the NCI CTCAE v5.0
Safety, tolerability and pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab (Adverse Events) [Biomarker part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Uncorrected QT interval, QTcF, PR duration, QRS interval and RR interval
From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks. | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Heart Rate
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Biomarker part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Maximum plasma concentration (Cmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Biomarker part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Time to reach maximum plasma drug concentration (Tmax) of ERY974
Pharmacokinetics of ERY974 in combination with atezolizumab and bevacizumab [Biomarker part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Time to reach maximum plasma drug concentration (AUC) of ERY974
Pharmacokinetics of ERY974 [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Maximum plasma concentration (Cmax) of ERY974
Pharmacokinetics of ERY974 [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Time to reach maximum plasma drug concentration (Tmax) of ERY974
Pharmacokinetics of ERY974 [Mono dose escalation part] | From first dose until 28 days after the last dose of study treatment, assessed up to about 52 weeks.
  Area under the concentration versus time curve (AUC) of ERY974
Biomarkers of ERY974 [Mono dose escalation part] | From screening to 6weeks
  GPC3 IHC staining
Biomarkers of ERY974 [Mono dose escalation part] | From screening to 6weeks
  Immune-related molecule IHC
Biomarkers of ERY974 [Mono dose escalation part] | From screening to 6weeks
  Gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (11):
- Japan (5):
  - Chiba University Hospital, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kindai University Hospital, Sayama, Osaka
  - National Cancer Center Hospital, Chuo Ku, Tokyo
- Taiwan (6):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).

REFERENCES:
- [Derived] Komatsu SI, Kayukawa Y, Miyazaki Y, Kaneko A, Ikegami H, Ishiguro T, Nakamura M, Frings W, Ono N, Sakata K, Fujii T, Kishishita S, Kitazawa T, Endo M, Sano Y. Determination of starting dose of the T cell-redirecting bispecific antibody ERY974 targeting glypican-3 in first-in-human clinical trial. Sci Rep. 2022 Jul 19;12(1):12312. doi: 10.1038/s41598-022-16564-x. PMID 35853994